CLINICAL TRIAL: NCT02748070
Title: The Role of Perioperative Systemic Steroids in Patients With Chronic Rhinosinusitis Without Polyps (CRSsNP)
Brief Title: Perioperative Oral Steroids for Chronic Rhinosinusitis Without Polyps (CRSsNP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Julia Noel, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 33096
Record Dates: First submitted 2016-04-15; First posted 2016-04-22 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Chronic Rhinosinusitis; Endoscopic Sinus Surgery; Chronic Rhinosinusitis Without Polyps; Oral Steroids
MeSH Terms: interventions — Prednisone; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Prednisone (Experimental): Provided oral steroid and topical steroid
  Interventions: Drug: Prednisone; Drug: Flonase
- Placebo (Placebo Comparator): Provided oral placebo and topical steroid
  Interventions: Drug: Flonase

INTERVENTIONS:
Drug: Prednisone
  Arms: Prednisone
Drug: Flonase

SUMMARY:
While oral steroids have been shown to be effective in the management of patients with chronic rhinosinusitis with polyps, its role in treating chronic rhinosinusitis without polyps (CRSsNP) is ambiguous. Despite a lack of strong clinical evidence to suggest a benefit in this disease state, steroids are often prescribed as a component of post-operative care after sinus surgery for patients without polyps. Oral steroids carry with them significant adverse effects, and should be prescribed thoughtfully. The aims of this study are to determine if oral steroids in the peri-operative period improves patient outcomes in CRS without polyps.

ELIGIBILITY:
Inclusion Criteria:

* CRSsNP as defined by Clinical Practice Guideline (Update) on Adult Sinusitis
* scheduled to undergo endoscopic sinus surgery

Exclusion Criteria:

* chronic rhinosinusitis with polyps (CRSwNP)
* Aspirin exacerbated respiratory disease
* Cystic fibrosis
* Immunosuppressive states (Human immunodeficiency virus, transplant)
* Oral steroid use within 30 days of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-08; Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia E Noel, MD, Principal Investigator — Stanford University; Michael T Chang, MD, Principal Investigator — Stanford University; Peter H Hwang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang MT, Noel J, Ayoub NF, Qian ZJ, Dholakia S, Nayak JV, Patel ZM, Hwang PH. Oral Corticosteroids Following Endoscopic Sinus Surgery for Chronic Rhinosinusitis Without Nasal Polyposis: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 May 1;147(5):434-441. doi: 10.1001/jamaoto.2021.0011. PMID 33662124

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisone: Participants received oral prednisone taper for 12 days postoperatively.
- Placebo: Participants received oral placebo for 12 days postoperatively.
Period: Overall Study
Arm/Group | Prednisone | Placebo
Started | 41 | 40
Randomized and Treated | 40 | 40
Completed | 33 | 39
Not Completed | 8 | 1

BASELINE CHARACTERISTICS:
Population: Patients who completed the protocol are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone | Placebo | Total
Number analyzed (Participants) | 33 | 39 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (15.3) | 49.9 (14.7) | 49.4 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 18 | 18 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30 | 30 | 60
  Black | 0 | 2 | 2
  Asian | 1 | 4 | 5
  Latino | 2 | 2 | 4
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 39 | 72
Sino-nasal Outcome Test 22 (SNOT-22) [Mean (Standard Deviation); unit: score on a scale] — SNOT-22 is a validated scale which measures sinonasal symptoms for sinusitis patients. The 22 questions are rated on a scale of 0-5 for a maximum total score of 110. Higher scores represent more symptomatic patients.
  score on a scale | 43.8 (21.5) | 43.0 (22.4) | 43.4 (21.8)
Lund-Kennedy Endoscopy Score [Mean (Standard Deviation); unit: score on a scale] — The Lund-Kennedy score is a validated scale by which clinicians grade the endoscopic appearance of the sinonasal cavity for sinusitis patients. There are 5 parameters rated on a scale of 0-2 for each side of the nose, for a maximum total score of 20 points. Higher scores represent a worse endoscopic appearance.
  score on a scale | 3.8 (3.1) | 2.9 (2.5) | 3.3 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Sino-nasal Outcome Test (SNOT-22) Over Time
Description: SNOT-22 is a validated scale which measures sinonasal symptoms for sinusitis patients. The 22 questions are rated on a scale of 0-5 for a maximum total score of 110. Higher scores represent more symptomatic patients.
Time Frame: Baseline, 1, week, 1 month, 3 months, and 6 months
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 33 | 39
score on a scale
  Baseline | 43.8 (21.5) | 42.9 (22.4)
  1 week | 39.7 (22.5) | 38.5 (21.2)
  1 month | 26.6 (20.8) | 28.6 (18.0)
  3 months | 28.3 (19.5) | 20.3 (15.2)
  6 months | 34.2 (20.6) | 25.2 (19.7)
Statistical Analysis 1: Comparison: Prednisone vs Placebo; Comparison of baseline and 1 week; Test type: Other; p = 0.819, t-test, 2 sided
Statistical Analysis 2: Comparison: Prednisone vs Placebo; Comparison of baseline and 1 month; Test type: Other; p = 0.665, t-test, 2 sided
Statistical Analysis 3: Comparison: Prednisone vs Placebo; Comparison of baseline and 3 months; Test type: Other; p = 0.071, t-test, 2 sided
Statistical Analysis 4: Comparison: Prednisone vs Placebo; Comparison of baseline and 6 months; Test type: Other; p = 0.097, t-test, 2 sided

2. Primary Outcome: Lund Kennedy Endoscopy Score Over Time
Description: The Lund-Kennedy score is a validated scale by which clinicians grade the endoscopic appearance of the sinonasal cavity for sinusitis patients. There are 5 parameters rated on a scale of 0-2 for each side of the nose, for a maximum total score of 20 points. Higher scores represent a worse endoscopic appearance.
Time Frame: Baseline, 1, week, 1 month, 3 months, and 6 months
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 33 | 39
score on a scale
  Baseline | 2.9 (2.5) | 3.8 (3.1)
  1 week | 5.9 (3.0) | 5.3 (2.6)
  1 month | 3.5 (2.7) | 3.8 (2.6)
  3 months | 1.9 (2.1) | 2.4 (2.1)
  6 months | 1.3 (1.7) | 1.8 (1.8)
Statistical Analysis 1: Comparison: Prednisone vs Placebo; Comparison of baseline and 1 week; Test type: Other; p = 0.376, t-test, 2 sided
Statistical Analysis 2: Comparison: Prednisone vs Placebo; Comparison of baseline and 1 month; Test type: Other; p = 0.685, t-test, 2 sided
Statistical Analysis 3: Comparison: Prednisone vs Placebo; Comparison of baseline and 3 months; Test type: Other; p = 0.388, t-test, 2 sided
Statistical Analysis 4: Comparison: Prednisone vs Placebo; Comparison of baseline and 6 months; Test type: Other; p = 0.233, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were collection as usual; additionally, a patient-completed survey was used to measure adverse effects related to treatment. This survey was designed to capture potential side effects of systemic corticosteroids.
Arm/Group | Prednisone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 14/41 | 19/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prednisone (N=41) | Placebo (N=40)
Easy bruising (Blood and lymphatic system disorders) | 0 | 3 — Collected by patient-completed survey
Water retention (Blood and lymphatic system disorders) | 3 | 4 — Collected by patient-completed survey
Blurry vision (Eye disorders) | 3 | 5 — Collected by patient-completed survey
Increased appetite (Gastrointestinal disorders) | 4 | 2 — Collected by patient-completed survey
Weight gain (Gastrointestinal disorders) | 2 | 4 — Collected by patient-completed survey
Stomach discomfort (Gastrointestinal disorders) | 8 | 11 — Collected by patient-completed survey
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 9 — Collected by patient-completed survey
Headache (Nervous system disorders) | 12 | 18 — Collected by patient-completed survey
Mood swings (Psychiatric disorders) | 3 | 4 — Collected by patient-completed survey
Increased aggression (Psychiatric disorders) | 1 | 2 — Collected by patient-completed survey
Nervouseness (Psychiatric disorders) | 6 | 5 — Collected by patient-completed survey
Difficulty sleeping (Psychiatric disorders) | 12 | 13 — Collected by patient-completed survey
High blood pressure (Vascular disorders) | 1 | 1 — Collected by patient-completed survey
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-02-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT02748070/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT02748070/SAP_001.pdf